CLINICAL TRIAL: NCT00002428
Title: A Phase I/II Safety and Immunogenicity Trial of UBI Microparticulate Monovalent (HIV-1 MN) Branched Peptide Vaccine in HIV-1 Seronegative Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Biomedical (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Prevention
Other Study IDs: 091; UBI V106
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1996-03

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; HIV-1; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: HIV-1 Peptide Vaccine, Microparticulate Monovalent
Biological: rgp120/HIV-1MN Monovalent Octameric V3 Peptide Vaccine

SUMMARY:
To evaluate the safety and immunogenicity of a combination of microparticulate monovalent HIV-1 MN synthetic branched peptide candidate vaccine for oral administration and monovalent HIV-1 MN synthetic branched peptide vaccine in alum for intramuscular administration in intermediate or higher risk HIV-negative volunteers.

DETAILED DESCRIPTION:
Volunteers receive one of two schedules of vaccines or placebo administered at days 0, 28, and 168. Specifically, group 1 receives oral microparticulate monovalent vaccine over 3 consecutive days on days 0, 1, and 2, and 28, 29, and 30, with the intramuscular monovalent vaccine given on day 168. Group 2 receives the intramuscular vaccine first, on day 0, followed by the oral form given on days 28, 29, and 30 and 168, 169, and 170. Volunteers are followed for 1 year.

ELIGIBILITY:
Inclusion Criteria

Volunteers must have:

* Normal history and physical exam.
* HIV negativity.
* CD4 count >= 400 cells/mm3.
* Intermediate or high risk sexual behavior or a history of injection drug use within 12 months prior to study entry.
* Normal urine dipstick with esterase and nitrite.

Exclusion Criteria

Co-existing Condition:

Volunteers with the following symptoms or conditions are excluded:

* Active tuberculosis.
* Occupational or other responsibilities that would prevent completion of study.

Volunteers with the following prior conditions are excluded:

* History of immunodeficiency, chronic illness, autoimmune disease, or use of immunosuppressive medications.
* Psychiatric, medical, or substance abuse problems within the past 6 months that would affect ability to participate in study.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* History of inflammatory gastrointestinal disease, celiac disease, or intestinal malignancy.
* Acute gastroenteritis or gastrointestinal surgery within the past 12 months.

Prior Medication:

Excluded:

* Live or attenuated vaccine within the past 60 days.
* Illicit or experimental agents within the past 30 days. Intermediate or high risk sexual behavior. Injection drug use within the past 12 months.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Univ of California at San Francisco Gen Hosp, San Francisco, California, United States

REFERENCES:
- [Background] Lambert JS, Keefer M, Mulligan MJ, Schwartz D, Mestecky J, Weinhold K, Smith C, Hsieh R, Moldoveanu Z, Fast P, Forrest B, Koff W. A Phase I safety and immunogenicity trial of UBI microparticulate monovalent HIV-1 MN oral peptide immunogen with parenteral boost in HIV-1 seronegative human subjects. Vaccine. 2001 Apr 30;19(23-24):3033-42. doi: 10.1016/s0264-410x(01)00051-2. PMID 11311997